CLINICAL TRIAL: NCT05920005
Title: A Multicenter, Double-blind, Controlled, Randomized Trial to Evaluate the Association Candesartan Cilexetil + Chlorthalidone + Amlodipine Versus Exforge HCT®️ for Systemic Arterial Hypertension
Brief Title: Candesartan Cilexetil + Chlorthalidone + Amlodipine Versus Exforge HCT®️ for Systemic Arterial Hypertension
Acronym: OPTION TREAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB2009
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Chlorthalidone; Amlodipine; Exforge HCT; Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: A multicenter, double-blind, phase III, parallel, controlled and randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experimental/comparator drug has different characteristics. To allow blinding, the Double-Dummy method will be performed, where study sites will receive two drug presentations (active and placebo), thus preventing any violation of blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Association of candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg (Experimental): The participant will take, once a day, 01 tablet of the active experimental drug (association candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg), plus 01 placebo, both orally.
  Interventions: Drug: candesartan cilexetil + chlorthalidone + amlodipine
- Exforge HCT® (valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg) (Active Comparator): The participant will take 01 tablet of Exforge HCT® active comparator (valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg) plus 01 placebo, both orally.
  Interventions: Drug: Exforge HCT® (valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg)

INTERVENTIONS:
Drug: candesartan cilexetil + chlorthalidone + amlodipine — Antihypertensive drugs in a single tablet (association candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg)
  Arms: Association of candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg
Drug: Exforge HCT® (valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg) — Antihypertensive drugs in a single tablet (association valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg)
  Arms: Exforge HCT® (valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg)

SUMMARY:
This study will evaluate the safety and efficacy of a new combination of 3 (three) antihypertensive drugs in a single pill (candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg) compared with another combination of 3 (three) antihypertensive drugs (Exforge HCT® [valsartan 160mg + hydrochlorothiazide 12.5mg + amlodipine 5mg]). This will be a non-inferiority trial and the primary outcome will be blood pressure control after 12 weeks of treatment.

DETAILED DESCRIPTION:
This phase III, multicenter, randomized, double-blind, controlled, parallel trial will evaluate the non-inferiority of the association between candesartan cilexetil 16mg + chlorthalidone 12.5mg + amlodipine 5mg in relation to Exforge HCT® (valsartan 160mg + hydrochlorothiazide 12 5mg + amlodipine 5mg) in the treatment of systemic arterial hypertension. A total of 698 participants will be included. Follow-up visits will occur four, eight, and twelve weeks after the date of the randomization visit. A telephone contact will be performed 30 days after the end of treatment. The primary efficacy outcome is the mean change in blood pressure, measured at the research site, 12 weeks after starting treatment, compared to baseline. Incidence of adverse events will be collected from the first dose of treatment up to 30 days after the end of the treatment foreseen in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged 18 years or older;
* Currently on dual antihypertensive therapy for at least 8 weeks, and non responders to that treatment, defined as measurements of SBP ≥ 140 mmHg and ≤180 mmHg and/or DBP≥90mmHg and ≤110 mmHg, assessed at the screening visit and randomization visit (both conditions are in accordance with the Brazilian Hypertension Guideline - 2020);
* Able to understand and consent to their participation in this clinical trial, manifested by signing the Informed Consent Form;

Exclusion Criteria:

* Any significant clinical condition that, in the investigator's opinion, may interfere with participant safety;
* Any laboratory test finding that, in the investigator's opinion, may interfere with participant safety;
* Suspected or diagnosed with COVID 19;
* History of hypersensitivity to components of drugs used during the trial or to drugs derived from sulfonamides;
* Pregnant or breastfeeding women;
* Women in a reproductive age who do not agree to use contraceptive methods;
* Male participants who do not agree to use contraceptive methods;
* Participation in clinical trial protocols in the last 12 (twelve) months, unless the investigator judges that there may be a direct benefit to the participant;
* Participant who has some kind of relationship up to the second degree or bond with collaborators or employees of the Sponsor and the Research site;
* Estimated glomerular filtration rate (eGFR) less than 45 ml/min /1.73m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) or end-stage renal disease;
* Severe liver dysfunction;
* Cardiogenic shock or reduced ejection fraction heart failure with a left ventricular ejection fraction less than or equal to 50%;
* Symptomatic congestive heart failure class II, III or IV, according to the New York Heart Association and/or participants with a history of infarction, unstable angina or cerebrovascular accident in the last 6 months prior to the beginning of the study;
* Clinically relevant ventricular cardiac arrhythmias;
* Obstructive coronary artery disease planning percutaneous or surgical intervention;
* Dementia syndrome;
* History of alcohol or illicit drug addiction in the six months prior to the date of signature of the Informed Consent Form;
* Obstructive biliary disorders;
* Refractory hypokalemia and/or conditions involving marked potassium loss, hyperkalemia (>5,5 mmol/L), and/or hyponatremia;
* History of symptomatic hyperuricemia;
* History of secondary hypertension;
* History of cancer, without documentation of remission/cure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure (SBP) | 12 weeks
  The primary efficacy endpoint is the mean change in systolic blood pressure, measured at the site, 12 weeks after starting treatment, compared to baseline.

SECONDARY OUTCOMES:
Mean change in diastolic blood pressure (DBP) | 12 weeks
  Variation in diastolic blood pressure 4, 6 and 12 weeks after starting treatment
Participants with blood pressure (SBP <140 and DBP<90 mmHg) | 12 weeks
  Proportion of participants who reach the target blood pressure (SBP <140 and DBP<90mmHg) 4, 8 and 12 weeks after starting treatment
Participants with SBP <120 mmHg | 12 weeks
  Proportion of participants who reach the target blood pressure of SBP <120 mmHg 4, 8 and 12 weeks after starting treatment
Participants with SBP <140 mmHg | 12 weeks
  Proportion of participants who reach target systolic blood pressure (SBP <140 mmHg) 4, 8 and 12 weeks after starting treatment
Participants with DBP<90 mmHg | 12 weeks
  Proportion of participants who reach the target diastolic blood pressure (DBP<90 mmHg) 4, 8 and 12 weeks after starting treatment
Participants with reduction greater than or equal to 20 mmHg in SBP | 12 weeks
  Proportion of participants who show a reduction greater than or equal to 20 mmHg in systolic blood pressure 4, 8 and 12 weeks after the start of treatment
Participants with reduction greater than or equal to 10 mmHg in DBP | 12 weeks
  Proportion of participants who have a reduction greater than or equal to 10 mmHg in diastolic blood pressure 4, 8 and 12 weeks after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Oliveira Guimarães, MD, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (22):
- Brazil (22):
  - Hospital de Urgência e Emergência de Rio Branco, Rio Branco, Acre
  - Centro de Pesquisas Clinicas Dr. Marco Mota (Centro Universitario Cesmac/ Hospital do Coração de Alagoas), Maceió, Alagoas
  - Centro de Pesquisas em Diabetes e Doenças Endócrino Metabólicas LTDA, Fortaleza, Ceará
  - Vitoria Clinical Research Institute LTDA, Vitória, Espírito Santo
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Hospital Universitário Joao de Barros Barreto - UFPA, Belém, Pará
  - Hospital 9 de Julho, São Paulo, Please Select
  - Hospital Universitário Pedro Ernesto/UERJ, Rio de Janeiro, Rio de Janeiro
  - Instituto Atena de Pesquisa Clinica LTDA, Natal, Rio Grande do Norte
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CMEP Centro Multidisciplinar de Ensino Especializado e Pesquisa Ltda, Joinville, Santa Catarina
  - Centro de Pesquisa Clínica do Coração, Aracaju, Sergipe
  - Hospital Universitário São Francisco de Assis, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - LOEMA - Instituto de Pesquisa Clinica & Consultores LTDA., Campinas, São Paulo
  - Indacor Serviços Médicos, Indaiatuba, São Paulo
  - CIPES Centro Internacional de Pesquisa Clínica LTDA, São José dos Campos, São Paulo
  - InCor - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, São Paulo, São Paulo
  - Associação Lar São Francisco de Assis na Providência de Deus, São Paulo, São Paulo
  - Hospital M'Boi Mirim, São Paulo, São Paulo
  - Clínica Cardiológica, Votuporanga, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Madrini V Jr, Tavares CAM, Albuquerque MTA, Silvestre OM, Felicio JS, Silveira FS, Hissa MN, Antunes MO, Mota-Gomes MA, Vidotti MH, Fuchs FD, Marcondes-Braga FG, Filho CRH, Troiani do Nascimento C, Bastos RA, Brandao AA, Cestario EES, Bortolotto LA, Castilho VC, Lapa MG, Magaton EAP, Fernandes PB, Albuquerque CSN, Silva LR, Berwanger O, Guimaraes PO. Efficacy and Safety of a Novel Triple Single-Pill for Uncontrolled Hypertension: The OPTION TREAT Trial. JACC Adv. 2025 Oct;4(10 Pt 2):102175. doi: 10.1016/j.jacadv.2025.102175. Epub 2025 Aug 29. PMID 40892621